CLINICAL TRIAL: NCT03727269
Title: Role Of Wii Fit Game Based Abdomino-Pelvic Training In Females With Urinary Incontinence
Brief Title: Wii Fit Game Based Abdomino-Pelvic Training In Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU Mizna Saleh
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Incontinence, Urinary
Keywords: Wii Fit; Urinary Incontinence; Females; Abdomino-Pelvic Training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Experimental group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wii Fit Training Experimental Group (Experimental): receiving Wii fit based abdomino-pelvic training
  Interventions: Other: Wii Fit Training Experimental Group
- Conventional Training Control Group (Active Comparator): receiving conventional pelvic floor exercises.
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Wii Fit Training Experimental Group — Experimental group receiving wii fit game based abdomino-pelvic training. A specific protocol was developed by the researchers. Wii fit games which promote exercises focusing on the abdominopelvic cavity strengthening, using as a therapeutic means a Wii™ console with a Wii Fit Plus™ CD game. The protocol was design that which playing games participant perform different pelvic movements such as anteversion, retroversion, lateral tilt and circumduction that maintain trunk control and stabilization with mild abdomino-pelvic muscle activation. Duration of each game is 5 minutes with 90 seconds interval between them twice a week. After performing the sequence of virtual games, a series of abdominopelvic and lower limb muscle stretching exercises will done.
  Arms: Wii Fit Training Experimental Group
Other: Conventional Training — Control group (n=20) receiving conventional pelvic floor exercises. Conventional exercises includes:
  1. Knack Maneuver (Ashton -Miller 1998, 2008)
  2. Pelvic floor strengthening: kegel Exercise.
  3. -Lumbo-Pelvic Stabilization Exercise.
  4. Functional Training/ PFM Contraction during ADL
  5. Correction of biomechanical/structural deformities
  Arms: Conventional Training Control Group

SUMMARY:
This study is aimed to determine the effect of Wii fit based abdomino-pelvic training on strength of pelvic floor muscles and on symptoms of urinary incontinence in females. An experimental, randomized controlled trial will be performed. Both reproductive and postmenopausal females with stress urinary incontinence will be included. 40 participants would be randomly distributed in experimental group (n=20) receiving wii fit based abdomino-pelvic training and control group (n=20) receiving conventional pelvic floor exercises. Pelvic floor strength would be assessed before and after by Digital method and EMG biofeedback. Urinary symptoms would be assessed by bladder diary, pad test and International consultation on Incontinence Questionnaires. Health related Quality of life questionnaire would also be used as an outcome measure. Data will be analyzed on SPSS 21 version using descriptive and inferential statistics

DETAILED DESCRIPTION:
Loss of bladder control results causes the accidental leak of urine is called urinary incontinence. It may be slightly bothersome or totally debilitating. It may leads to embarrassment and keeps them away from enjoying many physical activities, including exercising. Urinary incontinence may develop emotional distress because of some outside factors, such as difficulty getting to standing position or only being able to walk slowly, which prevent them from getting to the toilet on time.

Old women experience urinary incontinence more than young women or young girls. Muscles in the wall of bladder contracts during urination. Sphincter muscles surrounding the urethra relax which let the urine to pass out from the body. Incontinence will occur when the muscles of bladder suddenly contracts or are not strong enough to hold back the urine. Then the urine may escape with less pressure than usual when the muscles are damaged, this causing a change in the position of the bladder.

Stress incontinence is the most common type of urinary incontinence. 80% of the females suffering from urinary incontinence have stress urinary incontinence. Obese women having greater intra-abdominal pressure leads to weakening of pelvic floor muscle which causes stress incontinence.

During pregnancy, child birth and menopause physical changes results in the weakening of muscles of bladder. As the result of physical exertions, muscles of bladder become weak that increase intra-abdominal pressure leakage may cause. Leakage may occur during coughing, sneezing or heavy lifting.

Wii fit games are computer-generated scenario that simulates experience through senses and perception. This approach is being used by physical therapist so than their patient stick to their exercise protocol and it enhance their training and functional level. Wii fit game based pelvic floor muscle exercises helps the pelvic floor muscle to strengthen by different movements such as anteversion,, retroversion, lateral tilting, truck rotation, circumduction and pelvic stabilization. video game based treatment that enhance patients' motivation, functional training and hence adherence to exercise regimen. As clinical practice in women's health physical therapy lacks options for pelvic floor muscle training and wii fit game based pelvic floor rehabilitation is an innovated method so could be a valuable adjunct in management of female urinary incontinence protocol.

ELIGIBILITY:
Inclusion Criteria:

* • Females with only stress urinary incontinence (SUI).

Exclusion Criteria:

* Females with urinary tract infection.
* Females with myopathy, neurological abnormalities, cognitive or physical disorder that could hinder in training and assessment.
* Pelvic floor muscle strength 0 on Modified oxford grading scale and pelvic organ prolapse greater than or equal to 3 on pelvic organ Quantification (POP-Q) system.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal females
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
EMG biofeedback | 8 week
  EMG biofeedback device shows electrical activity of pelvic floor muscles and can assist with both muscle strengthening AND relaxation training

SECONDARY OUTCOMES:
Michigan Incontinence Symptoms Index: | 8th week
  Michigan incontinence symptoms index is a clinical measure of type, severity and bother related to urinary incontinence.The M-ISI is a parsimonious measure that has established reliability and validity on several levels and complements current clinical evaluative methods for patients with urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: imran Amjad, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood LN, Anger JT. Urinary incontinence in women. BMJ. 2014 Sep 15;349:g4531. doi: 10.1136/bmj.g4531. PMID 25225003
- [Background] Hilton P. Urinary incontinence in women. Br Med J (Clin Res Ed). 1987 Aug 15;295(6595):426-32. doi: 10.1136/bmj.295.6595.426. No abstract available. PMID 3115486
- [Background] Osborn DJ, Strain M, Gomelsky A, Rothschild J, Dmochowski R. Obesity and female stress urinary incontinence. Urology. 2013 Oct;82(4):759-63. doi: 10.1016/j.urology.2013.06.020. Epub 2013 Aug 22. PMID 23972338
- [Background] Burgio KL, Matthews KA, Engel BT. Prevalence, incidence and correlates of urinary incontinence in healthy, middle-aged women. J Urol. 1991 Nov;146(5):1255-9. doi: 10.1016/s0022-5347(17)38063-1. PMID 1942274
- [Background] Dobson HD, Pearl RK, Orsay CP, Rasmussen M, Evenhouse R, Ai Z, Blew G, Dech F, Edison MI, Silverstein JC, Abcarian H. Virtual reality: new method of teaching anorectal and pelvic floor anatomy. Dis Colon Rectum. 2003 Mar;46(3):349-52. doi: 10.1097/01.DCR.0000054639.29160.9E. PMID 12626910
- [Background] Martinho NM, Silva VR, Marques J, Carvalho LC, Iunes DH, Botelho S. The effects of training by virtual reality or gym ball on pelvic floor muscle strength in postmenopausal women: a randomized controlled trial. Braz J Phys Ther. 2016 Mar 22;20(3):248-57. doi: 10.1590/bjpt-rbf.2014.0148. PMID 27437716
- [Background] Botelho S, Martinho NM, Silva VR, Marques J, Carvalho LC, Riccetto C. Virtual reality: a proposal for pelvic floor muscle training. Int Urogynecol J. 2015 Nov;26(11):1709-12. doi: 10.1007/s00192-015-2698-5. Epub 2015 Apr 30. PMID 25925487
- [Background] Steenstrup B, Giralte F, Bakker E, Grise P. [Evaluation of the electromyography activity of pelvic floor muscle during postural exercises using the Wii Fit Plus(c). Analysis and perspectives in rehabilitation]. Prog Urol. 2014 Dec;24(17):1099-105. doi: 10.1016/j.purol.2014.09.046. Epub 2014 Oct 23. French. PMID 25450755
- [Background] Elliott V, de Bruin ED, Dumoulin C. Virtual reality rehabilitation as a treatment approach for older women with mixed urinary incontinence: a feasibility study. Neurourol Urodyn. 2015 Mar;34(3):236-43. doi: 10.1002/nau.22553. Epub 2014 Jan 10. PMID 24415577
- [Background] Bertotto A, Schvartzman R, Uchoa S, Wender MCO. Effect of electromyographic biofeedback as an add-on to pelvic floor muscle exercises on neuromuscular outcomes and quality of life in postmenopausal women with stress urinary incontinence: A randomized controlled trial. Neurourol Urodyn. 2017 Nov;36(8):2142-2147. doi: 10.1002/nau.23258. Epub 2017 May 16. PMID 28508398
- [Background] Capelini MV, Riccetto CL, Dambros M, Tamanini JT, Herrmann V, Muller V. Pelvic floor exercises with biofeedback for stress urinary incontinence. Int Braz J Urol. 2006 Jul-Aug;32(4):462-8; discussion 469. doi: 10.1590/s1677-55382006000400015. PMID 16953917
- [Background] Thubert T, Deffieux X, Jousse M, Guinet-Lacoste A, Ismael SS, Amarenco G. Influence of a distraction task on pelvic floor muscle contraction. Neurourol Urodyn. 2015 Feb;34(2):139-43. doi: 10.1002/nau.22524. Epub 2014 Feb 12. PMID 24519688
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322